CLINICAL TRIAL: NCT04245332
Title: Effects of Fish Oil Supplementation in Combination With Resistance Exercise Training on Body Composition, Strength and Neuromuscular Function in Young, Resistance-Trained Individuals: A Randomized, Open-Label, Placebo-Controlled Trial
Brief Title: Effects of Fish Oil and Resistance Training on Muscle Mass and Function
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 restrictions on research at University
Sponsor: Rowan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro2019000649
Record Dates: First submitted 2020-01-27; First posted 2020-01-28 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Fat-free Masss; Muscle Strength; Neuromuscular Function
MeSH Terms: interventions — Fish Oils; Coconut Oil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fish Oil (Experimental): This group will receive fish oil (4g/d).
  Interventions: Dietary Supplement: Fish oil
- Placebo (Placebo Comparator): This group will receive coconut oil (4g/d) as an iso-energetic, iso-lipidic placebo comparator to the fish oil arm.
  Interventions: Dietary Supplement: Coconut oil

INTERVENTIONS:
Dietary Supplement: Fish oil — Fish oil-derived omega-3 polyunsaturated fatty acids (4g fish oil concentrate: 2g EPA+ 1g DHA)
  Other Names: NOW Foods Ultra Omega-3
  Arms: Fish Oil
Dietary Supplement: Coconut oil — Coconut oil (4g/d)
  Other Names: NOW Foods Virgin Coconut Oil Softgels
  Arms: Placebo

SUMMARY:
This study consists of a free-living, 6-week fish oil (FO) or placebo (PLA) supplementation intervention alongside participants' habitual resistance exercise training (RET) regimens. Twenty young, healthy resistance-trained subjects who do not currently supplement with FO will be recruited to participate. An eligible participant will be between ages 18 and 35 and will have a minimum of two years of RET experience. Participants will be randomized into a FO group and a PLA group. The FO group will supplement with 4g/day of FO (4g fish oil concentrate: 2g EPA+ 1g DHA) and the PLA group will consume 4g/day of coconut oil (saturated fatty acids), as administered via gel capsules, in conjunction with their current RET program. Prior to intervention all participants will complete baseline biometric, strength, and neuromuscular testing. Participants will also have blood drawn to test for omega-3 fatty acid status, and complete and return a 3-day diet record and a physical activity recall. In order to monitor adherence to supplementation, FO and PLA bottles will also be returned weekly and pills will be counted. 3-day diet records will be obtained to ensure calorie and protein intakes remain consistent throughout the intervention period. Weekly physical activity records will also help to ensure consistency of participant training and to make sure all participants are following their training regimes in a progressive fashion. Following 6 weeks of FO or PLA supplementation, subjects will repeat all initial biometric, strength and neuromuscular testing, as well as a second, post-intervention blood draw.

DETAILED DESCRIPTION:
Potential participants will report to the Human Performance Lab (HPL) in James Hall to complete the screening process. They will complete the informed consent form process with a member of the research team before providing any protected health information (PHI). The screening process has two components: questionnaires and physical measures. Potential participants will complete the following questionnaires: Stanford 7-Day Physical Activity Questionnaire and a Medical History Questionnaire. Participants will complete the following physical measures: height, weight, waist and hip circumference, and blood pressure will be assessed and followed by calculations of body mass index (BMI) and waist to hip ratio (WHR). The final measure will be a determination of fasting total cholesterol and blood glucose measured via capillary blood from a finger prick using an automated analyzer. The purpose of the screening process is to determine if a participant is healthy and can safely participate in exercise testing, and to determine their eligibility to participate in the study based on the criteria listed elsewhere.

Participants who meet the eligibility criteria and are willing to participate will be enrolled in the study and randomly assigned to FO or PLA via block randomization methods. Enrolled participants will return to the HPL in the morning to complete a battery of biometric tests (described below) and will be given two logs to complete to collect baseline data: the Stanford 7-Day Physical Activity Questionnaire and a 3-day diet log. The purpose of the physical activity log is to determine their average level of physical activity and training program. The purpose of the 3-day diet log is to record their normal dietary intake and to provide practice for completing these logs as they will be completed on a weekly basis during the supplement intervention period.

Participants will have the following physical measures recorded: height, weight, waist and hip circumference, body composition, and blood pressure. Participants will then have their resting metabolic rate (RMR) measured by indirect calorimetry. In preparation for this test participants will be asked to complete an overnight fast of at least 9 hours, abstain from caffeine for 12 hours and abstain from exercise and alcohol for 24 hours. Participants will be brought to a quiet room and asked to lie in a supine position for 30 minutes of rest. They will then be fitted with a breathing mask connected to the metabolic cart and their breath will be analyzed for 15 minutes while they continue to lie in a supine position. Their total energy expenditure will be calculated using their RMR and a physical activity factor based on their level of physical activity obtained from the Stanford 7-Day Physical Activity Questionnaire. Subject's total daily calorie requirements will then be verified using their 3-day diet record and the Mifflin-St. Jeor prediction equation. In order to ensure that participants are consuming enough calories in order to maintain their body weight during the 6-week supplementation period, the research team will use the average of participant's total calorimetric data (based on RMR), 3-day diet log, and the Mifflin-St. Jeor estimate.

Participants will be sent pre-participation instructions before testing to ensure they arrive at the HPL with proper exercise attire and having abstained from caffeine for 12 hours and exercise and alcohol for 24 hours. They will report to the HPL to complete a 1RM test, a type of muscular strength assessment. This test will be performed for the back squat in a Smith machine with hand release breaks. Water will be provided and consumed ad libitum. Bench press and Squat will be completed with proper lifting technique as described by the National Strength and Conditioning Association (NSCA) guidelines.

Participants' lower body neuromuscular function, assessed via maximal voluntary contraction (MVC) and rate of force development (RFD), will be completed through the use of force transducers applied to the legs. Participants will be seated in a custom-made wooden box with a single axis transducer attached to one of its surfaces (SM-500, Interface Inc., Scottsdale, Arizona, USA). When subjects sit on the box, their knee and hip joints will be at approximately 70° and 90° of flexion from full extension, respectively. Subjects will be asked to cross their arms across their chest during the testing.

Dietary compliance will be monitored weekly during the free-living supplementation period using 3-day diet records and returned supplement pill bottles. 3-day diet records will be recorded by the participants and returned to the research team for analysis using professional nutrition analysis software (Food Processor, Oregon). Dietary analysis results will be discussed with the participant in order to help them adhere to dietary recommendations. Body weight measures will be recorded once per week to ensure a stable weight during the dietary intervention period. The participants will return supplement bottles weekly, and the research team will count and record any remaining capsules. Finally, physical activity logs will be collected every week to ensure diet and calorie recommendations are meeting the demands of RET.

ELIGIBILITY:
Inclusion Criteria:

* Young, healthy, resistance-trained men and women of all nationalities between the ages of 18-35

Exclusion Criteria:

* metabolic disease (diabetes or metabolic syndrome)
* cardiovascular disease
* pulmonary disease
* chronic inflammatory conditions (e.g. renal/kidney, liver, asthma, arthritis, autoimmune diseases, inflammatory bowel disease)
* neurological conditions (e.g. Parkinson's)
* sexually transmitted diseases
* cancer diagnosis within the previous 5 years
* currently smoking cigarettes
* hypertension
* hypercholesterolemia and/or dyslipidemia
* using medications to manage cholesterol, blood lipids, blood pressure, or diabetes
* taking performance-enhancing drugs and/or anabolic agents (e.g. testosterone, growth hormone, or beta-2 agonists)
* oral contraceptive use, are pregnant, or intend to become pregnant while enrolled in the study
* fish oil supplement use within the past 6 months
* fasting blood total cholesterol concentration >200mg/dl
* fasting blood glucose concentration >100mg/dl

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-29 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Total body fat-free mass (FFM) | 6 weeks
  Measured by bioelectrical impedance analysis (BIA)
Muscle strength | 6 weeks
  Measured by one-repetition maximal (1RM) strength in back squat, bench press, and knee extensor
Rate of force development (RFD) | 6 weeks
  Assessed by force transducers on legs and in hands
Maximal voluntary contraction (MVC) | 6 weeks
  Assessed by force transducers on legs and in hands

SECONDARY OUTCOMES:
Red blood cell omega-3 fatty acid concentrations (Eicosapentaenoic acid [EPA] and docosahexaenoic acid [DHA]) | 6 weeks
  Assessed by gas chromatography-mass spectrometry (GS-MS)

CONTACTS AND LOCATIONS:
Overall Officials: Dylan Klein, Ph.D., Principal Investigator — Rowan University
Locations (1):
- Rowan University, Glassboro, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No